CLINICAL TRIAL: NCT01170403
Title: Comprehensive Analyses of Multidetector-row Cardiac Computed Tomography Data of Over 15,000 Individuals in Korea
Brief Title: Comprehensive Analyses of Multidetector-row Cardiac Computed Tomography Data in Koreans
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: The Korean Society of Lipidology and Atherosclerosis (Unknown)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Other Study IDs: M10642140004-06N4214-00410
Record Dates: First submitted 2010-07-22; First posted 2010-07-27 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Coronary Disease
Keywords: coronary heart disease; Multidetector row cardiac computed tomography; type 2 diabetes; metabolic syndrome
MeSH Terms: conditions — Coronary Disease; Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NGT/IFG/DM, MeS/no-MeS: NGT: normal glucose tolerance IFG: impaired glucose tolerance DM : diabetes mellitus MeS: metabolic syndrome no-MeS: no metabolic syndrome

SUMMARY:
64 channel multidetector-row Computed Tomography (CT) has been introduced for use in the diagnosis of coronary heart disease. The investigators aimed to characterize coronary artery disease in type 2 diabetes mellitus and metabolic syndrome, and in particular plaque natures depending on different status of metabolic diseases. The investigators also aimed to analyze the risk factors associated with number and severity of stenosis as well as plaque characteristics using logistic regression models.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older

Exclusion Criteria:

* pregnant women
* patients with chronic kidney disease (Cr>2.0)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who had undertook a computed tomographic angiography (CTA) with 64-slice MDCT from January 2nd 2006 until August 21st 2008. Reasons for exam include screening in asymptomatic subjects, diagnosis in patients with angina pectoris, follow up after percutaneous coronary intervention or coronary artery bypass grafting, differential diagnosis in chest pain and so on.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2006-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Cardiovascular event | five years

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Bundang-gu, South Korea